CLINICAL TRIAL: NCT05998122
Title: Total Neoadjuvant Chemoradiotherapy Plus Anti-PD-1 in Subperitoneal High-Risk or Very High-Risk Patients With Locally Advanced Rectal Cancer: A Prospective, Single Arm, Exploratory Study
Brief Title: Total Neoadjuvant Chemoradiotherapy Plus Anti-PD-1 in Subperitoneal Patients With Locally Advanced Rectal CancerPatients With Locally Advanced Rectal Cancer: A Prospective, Single Arm, Exploratory Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Quan Wang, Prof., The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARS-RC06
Record Dates: First submitted 2023-08-11; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Locally Advanced Rectal Cancer; Total Neoadjuvant Treatment; Anti-PD-1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Radiation: Long-course chemoradiotherapy is delivered in 50 Gy/25 fractions with concurrent Capecitabine (825mg/m2, P.O. Bid, 5d/w).
  Drug: CapeOX (Capecitabine 1000mg/m2, P.O. Bid, d1-d14, q3w; Oxaliplatin 130mg/m2, i.v., d1, q3w), and Sintilimab (200mg, i.v. , d1).
  Surgical Approach: TME surgery, The surgical approach can be open, laparoscopic or robotic depending on the patient.
  Interventions: Other: nCRT → (CapeOX+Sintilimab)×6 → Surgery/W&W

INTERVENTIONS:
Other: nCRT → (CapeOX+Sintilimab)×6 → Surgery/W&W — Radiation: Long-course chemoradiotherapy is delivered in 50 Gy/25 fractions with concurrent Capecitabine (825mg/m2, P.O. Bid, 5d/w).
  Drug: CapeOX (Capecitabine 1000mg/m2, P.O. Bid, d1-d14, q3w; Oxaliplatin 130mg/m2, i.v., d1, q3w), and Sintilimab (200mg, i.v. , d1).
  Surgical Approach: TME surgery, The surgical approach can be open, laparoscopic or robotic depending on the patient.

SUMMARY:
Previously, preliminary results, from a subgroup analysis of STARS-RC03 (NCT04906044) conducted by our research team, showed that the 6-cycles consolidation chemotherapy combining with anti-PD-1 therapy had a better tumor regression advantage with a restricted safety profile contrasted with 3-cycle counterparts. Herein, we designed this study to further evaluate the short-term efficacy (such as pCR rate, R0 resection rate, etc.) and long-term survival (including DFS, OS, etc.) of 6-cycles consolidation therapy.

DETAILED DESCRIPTION:
The combination of total neoadjuvant treatment (TNT) and immunotherapy has shown a significant improvement in the pCR rate compared to the standard of care (SOC) or TNT alone for pMMR LARC. On this basis, we believe that this treatment mode will offers the opportunity of organ preservation for subperitoneal "Bad" or "Advanced" patients with LARC, who are initially assessed as unresectable or difficult to obtain R0 resection. Previously, preliminary results, from a subgroup analysis of STARS-RC03 (NCT04906044) conducted by our research team, showed that the 6-cycles consolidation chemotherapy combining with anti-PD-1 therapy had a better tumor regression advantage with a restricted safety profile contrasted with 3-cycle counterparts. Herein, we designed this study to further evaluate the short-term efficacy (such as pCR rate, R0 resection rate, etc.) and long-term survival (including DFS, OS, etc.) of 6-cycles consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The patients and their families are able to understand and are willing to participate in this clinical study, and sign an informed consent form.
2. Age: 18~75 years old, no gender limit;
3. Pathologically diagnosed rectal adenocarcinoma: differentiated into Grade 1-3, that is, high, medium, and poorly differentiated tubular adenocarcinoma; classified as pMMR/MSS.
4. The initial TNM risk category (from Rectal cancer: ESMO Clinical Practice Guidelines, 2017 edition) is as follows: 1) "Bad": cT3c/d or very low localisation levators threatened, MRF clear; cT3c/d mid-rectum, cN1-N2 (extranodal), EMVI+, limited cT4aN0; 2) "Advanced": cT3 with any MRF involved, any cT4a/b, lateral node+.
5. The lower edge of the tumor is located below the peritoneal reflex;
6. No distant transfer;
7. ECOG PS score 0-1 within 7 days before the first medication;
8. Hepatitis B Surface Antigen (HBsAg) (-) and Hepatitis B Core Antibody (HBcAb) (-). If HBsAg (+) or HBcAb (+), hepatitis B virus deoxyribonucleic acid (HBV-DNA) must be less than 1000 copies/mL or 200 IU/mL before entering the group.
9. HCV antibody (-)
10. The main organ function is normal.
11. No history of pelvic radiotherapy;
12. No history of rectal cancer surgery or chemotherapy;
13. Not accompanied by systemic infections requiring antibiotic treatment;
14. Heart, lung, liver, and kidney functions can tolerate surgery;
15. Others, based on the results of previous medical history, vital signs, physical examination or laboratory examination, the research doctor judges that you are suitable for participating in this clinical study.

Exclusion Criteria:

1. Recurrent rectal cancer;
2. Patients who are planning to undergo or have previously received organ or bone marrow transplantation;
3. Myocardial infarction or poorly controlled arrhythmia (including QTc interval ≥ 450 ms for males and ≥ 470 ms for females) occurred within 6 months before the first medication (QTc interval is calculated by Fridericia formula);
4. Existence of NYHA standard grade III to IV cardiac insufficiency or color Doppler ultrasound examination: LVEF (left ventricular ejection fraction) <50%;
5. Human immunodeficiency virus (HIV) infection;
6. Suffer from active tuberculosis;
7. Past and present patients with interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severely impaired lung function, etc., which may interfere with the detection and treatment of suspected drug-related lung toxicity;
8. Patients with active or suspicious autoimmune disease, or with a history of that;
9. Received treatment with live vaccines within 28 days before the first administration; except for inactivated viral vaccines for seasonal influenza;
10. Have received other antibody/drug treatments against immune checkpoints in the past, such as PD-1, PD-L1, CTLA4, etc.;
11. Known to have a history of severe allergies to any monoclonal antibody or research drug excipients;
12. In the past 5 years, patients have suffered from malignant tumors whose survival rate is significantly lower than the historical data of our rectal cancer survival rate (properly treated basal cell carcinoma, skin squamous cell carcinoma, small kidney cancer, breast cancer, and papillary thyroid carcinoma are not included here. range);
13. The patient has had arterial embolism diseases in the past 6 months, such as angina pectoris, MI, TIA, CVA, etc.;
14. Have received other types of anti-tumor or experimental treatments;
15. The patient is a female during pregnancy or lactation;
16. The patient has other diseases or abnormal mental states, which may affect the patient's participation in this study;
17. There are patients who may increase the risk of participating in research and research medication, or other severe, acute and chronic diseases, who are not suitable for clinical research based on the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CR) | Within one week after Last treatment
  defined as clinical complete response (cCR) or pathologic complete response (pCR) achieved after neoadjuvant therapy.

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) | 1/2/3 years from the date of receiving neoadjuvant therapy
  1/2/3 years disease-free survival
Recurrence -Free Survival (RFS) | 1/2/3 years from the date of receiving neoadjuvant therapy
  1/2/3 years recurrence -free survival
Overall Survival (OS) | 3 years from the date of receiving neoadjuvant therapy
  3 years overall survival
Local Recurrence (LR) Rate | 2 years from the date of receiving neoadjuvant therapy
  2-year local recurrence rate
Organ preservation rate | 1/2/3 years from the date of receiving neoadjuvant therapy
  Organ preservation rate
R0 Resection rate | Within one week after surgery
  R0 Resection rate
The incidence of serious adverse events | Within 3 months after Last medication
  Any treatment-related grade 3 or higher non-hematological adverse event determined by CTCAE version v 5.0.
QLQ-C30 score | up to 12 months
  Quality of Life Questionnaire C30
QLQ-C29 score | up to 12 months
  Quality of Life Questionnaire C29
Low Anterior Resection Syndrome (LARS) | up to 12 months
  Low Anterior Resection Syndrome Questionnaire
Quality of life and function assessment | up to 12 months
  IIEF-5 (international questionnaire of erectile function-5)score
Wexner score | up to 12 months
  Wexner incontinence score

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gu M, Guo Y, He L, Sun X, Liang T, Wang Z, Li Y, Liu Z, Wang J, Qiu X, Guo L, Chang P, Wang Q. Total neoadjuvant chemoradiotherapy plus anti PD-1 for mid-to-low locally advanced rectal cancer: study protocol of a prospective, single arm, phase II study (STARS - RC06). Front Oncol. 2025 Aug 8;15:1594927. doi: 10.3389/fonc.2025.1594927. eCollection 2025. PMID 40860797